CLINICAL TRIAL: NCT02424331
Title: Effect of Pursed Lips Breathing on Chest Wall, Mobility Diaphragmatic and Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Marcely Kellyane Florenço Barros, Master, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19309213.3.0000.5208
Record Dates: First submitted 2015-03-05; First posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Respiratory mechanics; Plethysmography; Diaphragm; Respiratory muscles; Breathing exercises
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quiet Breathing or Pursed Lips Breathing (Experimental): Free or natural breathing for six minutes.
  Interventions: Other: Pursed Lips Breathing; Other: Quiet Breathing

INTERVENTIONS:
Other: Pursed Lips Breathing — Pursed Lips Breathing for six minutes.
Other: Quiet Breathing

SUMMARY:
This study aimed to evaluate the acute effect of PLB technique on diaphragmatic mobility, the kinematics of the thoracoabdominal complex analysis of lung volumes and exercise tolerance in patients with Chronic Obstructive Pulmonary Disease (COPD). This is a study randomized cross-over clinical trial and blind, in subjects with Chronic Obstructive Pulmonary Disease (COPD) according to criteria of the Global Initiative for Chronic Obstructive Lung Disease (GOLD) (FEV1 / FVC <0.7 and FEV1 <80% predicted) selected at the Clinical Hospital of the Federal University of Pernambuco (UFPE) and Otavio de Freitas General Hospital (HGOF). The investigators recruited 13 patients COPD (according to previous sample calculation) aged between 40 and 80 years, of both sexes. The first day was held evaluation of lung function, respiratory muscle strength, body composition, dyspnea index and functional capacity. On the second day was held evaluation of thoracoabdominal complex kinematics by plethysmography Optoelectronics (OEP) with Quiet Breathing (QB) or pursed-lips breathing (PLB). Lung volumes with 2 minutes with QB and 6 minutes PLB or only 6 minutes by QB as randomization were observed. Before and after performing the requested breathing pattern diaphragmatic mobility was observed by Ultrasonography (US) and requested the patient an Inspiratory Capacity maneuver (IC). The evaluator who performed the ultrasound was blinded as to the beginning of the breathing pattern of order performed by the patient.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis with stage II-IV (GOLD),
* Stable clinical condition (no exacerbation or hospital admission in the last four weeks preceding the study)
* Absence of other disease that may potentially contribute to dyspnea (heart disease, congestive heart failure, neuromuscular diseases, severe postural changes)

Exclusion Criteria:

* BMI> 30 kg / m2
* Musculoskeletal limitations
* Use of oxygen therapy
* Extreme discomfort during the procedure application

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Chest wall (Analysis of lung volumes) | One day during eight minutes
  (L) by plethysmography optoelectronics.
Mobility diaphragmatic (mobility diaphragmatic (mm) by Ultrassonography) | One day, before and after eight minutes of pursed lips breathing
  Analysis of mobility diaphragmatic (mm) by Ultrassonography.
Exercise tolerance (Glittre AVD-Test) | One day, for six minutes approximately. The test will be repeated after 20 minutes of rest.
  Analysis by Glittre AVD-Test (capacity functional test) observing the test execution time (s).

SECONDARY OUTCOMES:
Dyspnea (Borg and MRC Scale) | One day, before and after implementation of Glittre-ADL Test
  Assessed by Borg and MRC Scale (Medical Research Council).

CONTACTS AND LOCATIONS:
Overall Officials: Armele D Andrade, Dra, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Clinical Hospital, Recife, Pernambuco, Brazil